CLINICAL TRIAL: NCT03217604
Title: A Phase 1, Randomized, Double-blind, Sponsor-open, Placebo-controlled, First-in-human Study To Evaluate The Safety, Tolerability, And Pharmacokinetics Of Single Ascending Oral Doses Of Pf-06852231 Administered To Healthy Adult Subjects
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single Doses of PF-06852231 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: C2561001; 2017-000799-26 (EudraCT Number)
Record Dates: First submitted 2017-07-06; First posted 2017-07-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
Keywords: PF-06852231; Safety; Tolerability; Pharmacokinetics; First-in-human; Healthy subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- PF-06852231 (Experimental): Single ascending doses of PF-06852231
  Interventions: Drug: PF-06852231

INTERVENTIONS:
Drug: Placebo — Treatment with placebo
  Arms: Placebo
Drug: PF-06852231 — Treatment with PF-06852231
  Arms: PF-06852231

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of single ascending doses of PF-06852231 after first-time administration to healthy adult subjects. The safety, tolerability, and pharmacokinetics of an active metabolite (PF-06892787) will also be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects of non-childbearing potential and male subjects, who at the time of screening are between ages of 18 and 55 years inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead electrocardiogram, or clinical laboratory tests.
2. Body mass index of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
3. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product (whichever is longer).
3. Screening supine BP greater than or equal to 140 mm Hg (systolic) or greater than or equal to 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is greater than or equal to 140 mm Hg (systolic) or greater than or equal to 90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility.
4. Screening supine 12-lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
5. Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level greater than or equal to 1.5x upper limit of normal (ULN);
   * Total bilirubin level greater than or equal to 1.5x ULN; subjects with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is less than or equal to ULN.
6. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
7. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
8. Other acute or chronic medical or psychiatric conditions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-07-13 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 14 days after last dose of study medication
  Treatment-related AE are any untoward medical occurrence attributed to study drug in a participant who received study drug. Treatment-emergent are events between first dose of study drug and up to Y days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to study drug is assessed either yes or no by the investigator. Participants with multiple occurrences of an AE within a category are counted once within the category.
Number of Participants With Laboratory Abnormalities | Baseline up to 14 days after last dose of study medication
  Following parameters were analyzed for laboratory examination: hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid albumin, total protein); urinalysis (decimal logarithm of reciprocal of hydrogen ion activity [pH], glucose, protein, blood, ketones, microscopy[if urine tested positive for blood or protein]).
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | 0, 1, 2, 4, 8, 12, 24, 48, 72 hours(h) post-dose
  Following parameters were analyzed for examination of vital signs: systolic and diastolic blood pressure, pulse rate, and body temperature.
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Findings | 0, 1, 2, 4, 8, 12, 24, 48, 72 h post-dose
  Absolute values and changes from baseline for ECG parameters
Abnormal rhythms as observed continuous cardiac telemetry | 8 h post-dose
  Cardiac rhythms measured by continuous cardiac monitoring

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for PF-06852231 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 h post-dose
  Maximum Observed Plasma Concentration (Cmax) for PF-06852231
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06852231 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 h post-dose
  Time to Reach Maximum Observed PF-06852231 Plasma Concentration (Tmax)
Area Under the Curve From Time Zero to Time of Last Measurable Plasma Concentration (AUClast) for PF-06852231 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 h post-dose
  AUClast = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to time of last measurable plasma concentration.
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for PF-06852231 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 h post-dose
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Plasma Decay Half-Life (t1/2) of PF-06852231 | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 h post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Maximum Observed Plasma Concentration (Cmax) for PF-06892787 (metabolite of PF-06852231) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 h post-dose
  Maximum Observed Plasma Concentration (Cmax) for PF-06892787
Time to Reach Maximum Observed Plasma Concentration (Tmax) for PF-06892787 (metabolite of PF-06852231) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 h post-dose
  Time to Reach Maximum Observed PF-06892787 Plasma Concentration (Tmax)
Area Under the Curve From Time Zero to Time of Last Measurable Plasma Concentration (AUClast) for PF-06892787 (metabolite of PF-06852231) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 h post-dose
  AUClast = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to time of last measurable plasma concentration.
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) for PF-06892787 (metabolite of PF-06852231) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 h post-dose
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Plasma Decay Half-Life (t1/2) of PF-06892787 (metabolite of PF-06852231) | 0, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48, 72 h post-dose
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C2561001&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Sponsor-open%2C+Placebo-controlled%2C+First-in-human+Study+To+Evaluate+The+Safety%2C+Tolerability%2C+And+Pharmacokinetics+Of+Single+Ascending+Oral+Doses+Of+Pf-06852231+Administered+To+Healthy+Adult+Subjects